CLINICAL TRIAL: NCT05526482
Title: Applicability of Respiratory Tele-physiotherapy in the Preoperative Context of Thoracic Surgery at the Hospital de la Santa Creu y Sant Pau (HSCSP).
Brief Title: Preoperative Treatment of Respiratory Physiotherapy in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TFR-2021-126
Record Dates: First submitted 2022-03-02; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Lung Cancer; Physical Therapy; Thoracic Surgery; Preoperative
Keywords: lung cancer; tele-physiotherapy; preoperative; thoracic surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: mobile app — preoperative respiratory exercises and thoracic surgery with a mobile application

SUMMARY:
The home confinement caused by the COVID-19 pandemic has aroused the need to use telematic communication systems to provide remote treatments. More and more research is being done on preoperative respiratory physiotherapy in patients undergoing thoracic surgery with lung cancer. It is a treatment that has great relevance in the prevention of postoperative complications and in the quality of life of the patient. Therefore, this study is proposed to highlight the applicability of a telematic system of preoperative physiotherapy treatment with the FISSIOS application at the Hospital de la Santa Creu i Sant Pau (HSCSP).

DETAILED DESCRIPTION:
A pilot cohort follow-up study is proposed based on the viability of a tele-physiotherapy program preoperative respiratory thoracic surgery for pulmonary cancer. The Patient selection will be done over a period of 2 months between January and February 2022, without participant limit during this period. The patient will have two face-to-face visits where the assessments and data will be collected. During follow-up patients will do 3-4 video conferencing with the principal investigator. For 3-4 weeks the patients will use the FISSIOS App to follow up of the exercises every day. The study will be conducted at the HSCSP in Barcelona. The results will be analyzed by the Epidemiology of the Hospital de Sant Pau

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-> 80 years. Candidates for CP resection with curative intent, either for VATS or thoracotomy, which meet the ppo-DLCO> 35% and ppo-FEV1> 35% surgical criteria, who agree to participate and sign the informed consent

Exclusion Criteria:

* Patients undergoing tumor resection for cancer requiring pneumonectomy, with cognitive impairment, which are outside the area of influence of the HSCSP or which do not have from an Android / iPhone Operating System (iOS) device. It is also considered an exclusion criterion not fulfilling 50% of the predefined time of the program (a week and a half) and surgical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is aimed at patients diagnosed with pulmonary cancer candidates for surgery with curative intent a the HSCSP.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Feability to implement a respiratory tele-physiotherapy program in patients diagnosed with Cancer Pulmonary candidates for thoracotomy or VATS at the Hospital de la Santa Creu i Sant Pau. | 1-4 weeks
  will be assessed over time of treatment. 80% compliance with treatment.

SECONDARY OUTCOMES:
Adherence with treatment time -minutes of treatment | 1-4 weeks
  we will collect them with the minutes of treatment that appear in the application
The capacity of effort- 6MWT (6 meters walking test) | 1-4 weeks
  the capacity of effort with the 6 minutes walking test Evaluate the capacity of effort before and after the tele-physiotherapy program in patients undergoing thoracic surgery diagnosed with lung cancer
Dyspnea- mMRC (modified Medical Research Council) | 1-4 weeks
  Dyspnea in activities of daily living before and after the program with mMRC. 0 Absence of dyspnea on intense exercise
  1 Dyspnea when walking fast on level ground, or when walking up a slight incline. pronounced. two Dyspnea causes you to be unable to keep up with other people in the same age walking on level ground or having to stop to rest when walking on level ground at your own pace. 3 Dyspnea makes you have to stop to rest after walking 100 meters or a few minutes after walking on the flat. 4 Dyspnea prevents the patient from leaving the house or appears with activities such as dressing or undress. tele-physiotherapy performed on patients diagnosed with CP who are candidates for surgery thoracic.
Quality of Life Questionnaire module for Lung Cancer patients QLQ-C30 | 1-4 weeks
  the evolution of health-related quality of life before and after the program with EORTC QLQ-C30.
  Quality of Life Questionnaire module for Lung Cancer patients QLQ-C30: All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  QLQ-LC 13: All of the scales and single item measures range in score from 0 to 100. A high score for the symptom scales / single items represents a high level of symptomatology or problems.
Quality of Life Questionnaire module for Lung Cancer patients QLQ-LC 13 | 1-4 weeks
  the evolution of health-related quality of life before and after the program with Quality of Life Questionnaire module for Lung Cancer patientsQLQ-LC 13.
  QLQ-LC 13: All of the scales and single item measures range in score from 0 to 100. A high score for the symptom scales / single items represents a high level of symptomatology or problems.
Anxiety and depression | 1-4 weeks
  the evolution of the degree of anxiety and depression before and after of the program.
  Each question is scored from 0-3. There are 14 questions of which 7 assess depression and 7 assess anxiety. Scoring: 0-7 Normal, 8-10 Borderline abnormal (borderline case), 11-21 Abnormal (case).
degree of satisfaction- satisfaction questionnaire | 1-4 weeks
  the degree of satisfaction of the program after the program. There are 2 closed questions and a question and a satisfaction rating of 0-10. 0 is the minimum satisfaction and 10 is the maximum satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Dolça Gras Pacheco, Msc, Principal Investigator — Col·legi de Fisioterapeutes de Catalunya
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain